CLINICAL TRIAL: NCT00181571
Title: A Double-Blind Comparison of Concerta and Placebo in Adults With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-p-000037
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: ADHD
Keywords: ADHD; Adults; Concerta; Double-Blind
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Concerta
  Interventions: Drug: methylphenidate HCl (Concerta)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: methylphenidate HCl (Concerta) — up to a maximum dose of 1.3 mg Concerta/kg/day, and not more than 144 mg/day for any subject regardless of weight.
  Other Names: Concerta
  Arms: 1
Drug: Placebo — up to a maximum dose of 1.3 mg Placebo /kg/day, and not more than 144 mg/day for any subject regardless of weight.
  Arms: 2

SUMMARY:
This is a double-blind, placebo-controlled study using daily doses of up to 1.3 mg/kg/day of Concerta in the treatment of adults with the DSM-IV diagnosis of attention deficit hyperactivity disorder (ADHD) (childhood onset). We hypothesize ADHD symptomatology in adults with DSM-IV ADHD will be responsive to Concerta treatment and Concerta-associated response of ADHD symptomatology in adults will be sustained over time.

DETAILED DESCRIPTION:
Concerta was specially developed to replace three-times-a-day IR methylphenidate, making it an ideal option for patients with ADHD. Moreover, the once-a-day administration of Concerta secures a steady delivery of methylphenidate across the day, minimizing the well-known risks of peaks and valleys of IR methylphenidate, which could offer an added advantage to the pharmacokinetic advantage of once-a-day administration. Despite these putative advantages, whether this new delivery system will lead to the same results as those documented with immediate-response methylphenidate in the treatments of adults with ADHD requires empirical corroboration. To this end we are conducting a randomized controlled clinical trial to evaluate the short- and medium-term safety and efficacy of Concerta in the treatment of adults with ADHD with and without co-morbid psychiatric disorders. We also wish to examine the role of genetics in predicting ADHD treatment response to Concerta. There is growing literature that supports the role of genetic factors in treatment response in youth with ADHD, and we seek to further explore this relationship in adults.

The proposed study includes the use of a 34-week design to document the response rate, assessment of the impact of Concerta on functional capacities (quality of life, psychosocial function) and cognition, and careful assessment of safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female outpatients older than 18 and younger than 55 years of age.
2. Subjects with the diagnosis of attention deficit hyperactivity disorder (ADHD), by DSM-IV, as manifested in clinical evaluation and confirmed by structured interview.
3. ADHD Symptom Checklist score > 24.
4. Patients with past history of depression, bipolar disorder, anxiety disorder (including OCD) without current disorder for > 3 months as ascertained through structured diagnostic interview and clinical exam.
5. Subjects treated for anxiety disorders and depression who are on a stable medication regimen for at least three months, and who have a disorder-specific CGI-Severity score ≤ 3 (mildly ill) and who have a score on the Hamilton-Depression and Hamilton-Anxiety rating scales below 15 (mild range).
6. Subjects with a past history of tics but tic free for > 1 year.
7. Subjects with past history of substance use disorders but substance free for > 6 months.
8. Subjects receiving non-MAOI antidepressants (e.g., SSRI's, bupropion, venlafaxine) or benzodiazepines who have been on a stable regimen for > 3 months for any of the conditions listed above.

Exclusion Criteria:

1. Any clinically unstable psychiatric conditions including the following: acute psychosis, acute panic, acute OCD, acute mania, acute suicidality, bipolar disorder, acute substance use disorders (alcohol or drugs, sociopathy, criminality, or delinquency.
2. Any metabolic, neurological, hepatic, renal, cardiovascular, hematological, opthalmic, or endocrine disease.
3. Clinically significant abnormal baseline laboratory values which include the following:

   1. Values > 20% above the upper range of the laboratory standard of a basic metabolic screen.
   2. Exclusionary blood pressure > 140 (systolic) and 90 (diastolic).
   3. Exclusionary ECG parameters: QTC > 460 msec, QRS > 120 msec, and PR > 200 msec. Subjects having ECG evidence of ischemia or arrhythmia as reviewed by an independent cardiologist.
4. Mental retardation (IQ <75).
5. Organic brain disorders.
6. Seizures or tics in the last year.
7. Pregnant or nursing females.
8. Subjects with current adequate treatment for ADHD or a history of a previous adequate trial of Concerta.
9. Non-English speaking subjects will not be allowed into the study for the following reasons:

   1. the assessment instruments are unavailable and have not been adequately standardized in other languages;
   2. our clinical trials facility is located in Cambridge and not at the MGH main campus; thus translators are unavailable;
   3. even if such translation services were available, the assessments in the English language conducted by English-speaking clinicians and raters with English-speaking subjects are already extremely time-consuming, lasting many hours, making it unfeasible, unrealistic, and of dubious clinical validity to conduct them with a translator with non-English-speaking subjects;
   4. psychiatric questionnaires and evaluations are taxing, and adding the complexity of a translator has the potential to make the patient experience even more exhausting

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 297 (Actual)
Dates: Start 2003-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Symptom reduction using ADHD-Clinical Global Impression and ADHD Symptom Checklist Severity scale administered at each visit. | 34 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Biederman J, Mick E, Fried R, Wilner N, Spencer TJ, Faraone SV. Are stimulants effective in the treatment of executive function deficits? Results from a randomized double blind study of OROS-methylphenidate in adults with ADHD. Eur Neuropsychopharmacol. 2011 Jul;21(7):508-15. doi: 10.1016/j.euroneuro.2010.11.005. Epub 2011 Mar 9. PMID 21303732